CLINICAL TRIAL: NCT01957501
Title: Detecting Depression and Bipolar Disorder in Adolescents Using a Biomarker Panel
Status: Terminated | Type: Observational
Why Stopped: Funding has been terminated for this study.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Kondo, MD, MD, University of Utah
Other Study IDs: Ridge II
Record Dates: First submitted 2013-09-10; First posted 2013-10-08 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Serum Biomarkers
Keywords: Major Depressive Disorder; Bipolar Disorder; Adolescents; Biomarker
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Major Depressive Disorder Participants
  Interventions: Other: MDDScoreTM
- Bipolar Disorder Participants:
  Interventions: Other: MDDScoreTM
- Healthy Control Participants
  Interventions: Other: MDDScoreTM

INTERVENTIONS:
Other: MDDScoreTM — The child will receive a single blood draw (about 10 mL).

SUMMARY:
Depression and bipolar disorder are major public health concerns for adolescents today. Teenage depression and bipolar disorder are associated with social isolation, family stress, school failure, substance abuse and suicide. Screening for depression and bipolar disorder so that treatment can be started early in the course of illness is an urgent public health priority. Many teens with bipolar disorder are incorrectly diagnosed as having unipolar depression. It is critical that adolescents receive proper screening and assessment that leads to an accurate diagnosis and treatment. An efficient, cost-effective, blood-based screening program could be performed on an annual or semi-annual basis to potentially detect depression and then differentiate between unipolar and bipolar depression. If this type of screening were able to detect a significant percentage of teens with depression or bipolar disorder, the positive impact on U.S. public health would be substantial. The purpose of this study is to conduct a pilot study to assess the probability of detecting adolescent unipolar and bipolar depression through blood samples.

ELIGIBILITY:
Inclusion of Major Depressive Disorder Participants:

1. Male and female patients between the ages of 13 and 17 years
2. Participants must be able to give informed assent, and parent(s)/guardian(s) must be able to give informed permission for study participation
3. Diagnosis of MDD or depression not otherwise specified, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-TR criteria (DSM-IV-TR)
4. Current mood state depressed for > 2 weeks

Inclusion of Bipolar Disorder Participants:

1. Male and female patients between the ages of 13 and 17 years
2. Participants must be able to give informed assent, and parent (s)/guardian (s) must be able to give informed permission for study participation
3. Diagnosis of Bipolar I Disorder, Bipolar II Disorder, or not otherwise specified, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-TR criteria
4. Current mood state depressed for > 2 weeks

Inclusion of Healthy Control Participants:

1. Males and females between the ages of 13 and 17 years
2. Participants must not meet DSM-IV-TR diagnostic criteria for a psychiatric or substance abuse disorder
3. Participants must be able to give informed assent and parent (s)/guardian (s) must be able to give informed permission for study participation

Exclusion Criteria:

Exclusion of Major Depressive Disorder and Bipolar Disorder Participants:

1. Meet the DSM-IV criteria for substance abuse or dependence in the last month
2. History of fainting or other significant adverse event during blood draws in the past
3. Dysthymia
4. Daily use of oral or inhaled steroids
5. High risk of suicidal behaviors, homicidal behaviors, or self-harm
6. A medical condition, such as Addison's Disease, which is highly likely to influence the inflammatory or HPA responses

Exclusion of Healthy Control Participants:

1. Clinically significant psychiatric or substance abuse disorder
2. Unstable medical or neurological illness
3. History of fainting or other significant adverse event during blood draws in the past
4. Daily use of oral or inhaled steroids
5. A medical condition, such as Addison's Disease, which is highly likely to influence the inflammatory or HPA responses

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants who respond to recruitment flyers displayed within the community.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Biomarker for Major Depressive Disorder (MDD) and Bipolar Disorder in Adolescents | 4 years
  The MDDScore™ will determine the biomarker of Major Depressive Disorder (MDD) and Bipolar Disorder. The MDDScore™ is determined using nine blood based biomarkers (inflammatory markers [4], stress related hormones [2], neuroendocrine [1] and metabolic proteins [2]) on physiological pathways related to MDD. The test results for the MDDScore™ range from 1 to 10. If the patient's score is 1, the patient has a less than 10% likelihood of having MDD. If the patient's MDDScore™ is 10, the patient has a greater than 90% likelihood of having MDD. An MDDScore™ of 5 or less is considered normal or negative and a score of 6 or more is considered "diseased" or positive. This same scoring system would hold true for classifying the likelihood of having bipolar disorder, as well. Test characteristics, such as sensitivity and specificity, are calculated based on this determination.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kondo, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Greden JF. The burden of disease for treatment-resistant depression. J Clin Psychiatry. 2001;62 Suppl 16:26-31. PMID 11480881
- [Background] Kendler KS, Karkowski LM, Prescott CA. Causal relationship between stressful life events and the onset of major depression. Am J Psychiatry. 1999 Jun;156(6):837-41. doi: 10.1176/ajp.156.6.837. PMID 10360120
- [Background] McEwen BS. Effects of adverse experiences for brain structure and function. Biol Psychiatry. 2000 Oct 15;48(8):721-31. doi: 10.1016/s0006-3223(00)00964-1. PMID 11063969
- [Background] Shelton RC. The molecular neurobiology of depression. Psychiatr Clin North Am. 2007 Mar;30(1):1-11. doi: 10.1016/j.psc.2006.12.005. PMID 17362799
- [Background] Pillay SS, Renshaw PF, Bonello CM, Lafer BC, Fava M, Yurgelun-Todd D. A quantitative magnetic resonance imaging study of caudate and lenticular nucleus gray matter volume in primary unipolar major depression: relationship to treatment response and clinical severity. Psychiatry Res. 1998 Dec 14;84(2-3):61-74. doi: 10.1016/s0925-4927(98)00048-1. PMID 10710164
- [Background] Iosifescu DV, Papakostas GI, Lyoo IK, Lee HK, Renshaw PF, Alpert JE, Nierenberg A, Fava M. Brain MRI white matter hyperintensities and one-carbon cycle metabolism in non-geriatric outpatients with major depressive disorder (Part I). Psychiatry Res. 2005 Dec 30;140(3):291-9. doi: 10.1016/j.pscychresns.2005.09.003. PMID 16298109
- [Background] Renshaw, PF, Bilello, JA , Pi, B. Multianalyte Biomarker Blood Test to Aid in Diagnosis,Treatment and Management of Major Depressive Disorder. Poster NR7-014, American Psychiatric Association Meeting, May 2009.
- [Background] Murray, CJL, Lopez, AD (Eds), The Global Burden of Disease, Cambridge Mass., Harvard University Press, 1996.
- [Background] Robins LN, Regier DA (Eds). Psychiatric Disorders in America, The Epidemiologic Catchment Area Study, 1990; New York: The Free Press. Items 1 - 20 of 204